CLINICAL TRIAL: NCT02493530
Title: A Phase 1 Dose Escalation and Expansion Study of TGR-1202 + Ruxolitinib in Subjects With Primary Myelofibrosis (PMF), Post-Polycythemia Vera MF (PPV-MF), Post-Essential Thrombocythemia MF (PET-MF), MDS/MPN, or Polycythemia Vera Resistant to Hydroxyurea
Brief Title: TGR-1202 + Ruxolitinib PMF PPV-MF PET-MF MDS/MPN Polycythemia Vera Resistant to Hydroxyurea
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Responsible Party: Principal Investigator, Michael Savona, Professor of Medicine; Director, Hematology Early Therapeutics Program, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC HEM 1538
Record Dates: First submitted 2015-07-01; First posted 2015-07-09 (Estimated); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Myelofibrosis; Polycythemia Vera
Keywords: MDS/MPN
MeSH Terms: conditions — Primary Myelofibrosis; Polycythemia Vera | interventions — umbralisib; ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Escalation and expansion (Experimental): TGR1202 and Ruxolitinib combination
  Interventions: Drug: TGR-1202; Drug: ruxolitinib

INTERVENTIONS:
Drug: TGR-1202 — Stage 1 will include myelofibrosis or hydroxyurea-resistant/refractory PV patients already taking therapeutic levels of ruxolitinib, but who are not achieving maximal response at highest tolerated dose of ruxolitinib.
  Stage 2 will include myelofibrosis or hydroxyurea-resistant/refractory PV patients who have never been on JAK-STAT inhibitory agents, and includes simultaneously initiation of both ruxolitinib and TGR-1202. TGR-1202 will be administered at or below the recommended dose established in Stage 1.
  Expansion will commence after proper combination doses of both agents is established.
Drug: ruxolitinib
  Other Names: Jakafi

SUMMARY:
This is a Phase 1, open-label, study of TGR-1202, a PI3K delta inhibitor, administered together with ruxolitinib in patients with myeloproliferative neoplasms (specifically: polycythemia vera, primary myelofibrosis, PPV-MF or PET-MF) and MDS/MPN.

DETAILED DESCRIPTION:
The escalation will include 2 initial sequential stages. Stage 1 will include myelofibrosis or hydroxyurea-resistant/refractory PV patients already taking therapeutic levels of ruxolitinib, but who are not achieving maximal response at the highest tolerated dose of ruxolitinib as discussed among investigators. Only TGR-1202 will be escalated in a modified 3+3 dose escalation algorithm to determine the MTD of TGR-1202 to be given with any given dose of ruxolitinib.

Stage 2 will include myelofibrosis or hydroxyurea-resistant/refractory PV patients who have never been on JAK-STAT inhibitory agents, and includes simultaneously initiation of both ruxolitinib and TGR-1202. In Stage 2, JAK Inhibitor naïve patients will receive TGR-1202 at the recommended dose established in Cohort 1, and ruxolitinib. As patients in Stage 1 will be on ruxolitinib at different doses, dose levels in Stage 2 will expand to meet requirements for safety analysis.

ELIGIBILITY:
Inclusion Criteria:

* Must voluntarily sign an ICF; and must be able to meet all study requirements
* For escalation, subjects must have a pathologically confirmed diagnosis of PPV-MF, PETMF, or PMF as per the EHA or WHO diagnostic criteria (note that all diagnoses must include the presence of at least Grade 1 marrow fibrosis according to the European Consensus on Grading of BM Fibrosis as well as int-1, int-2, or high risk disease according to the IWG-MRT Dynamic IPSS; Patients with PV may enter the trial if they meet the labeled indication for ruxolitinib (eg hydroxyurea resistant or refractory);

  * Escalation Stage 1 patients: who have not achieved normalization of splenomegaly, symptomology, or blood counts with at least 8 weeks therapy with a steady dose of ruxolitinib
  * Escalation Stage 2: patients who have not yet received therapy with any JAK-STAT inhibitory agents or patients on at least 8 weeks of a steady dose of ruxolitinib; patients with exposure to other JAK-STAT inhibitory agents are not eligible. After discussion with the study chair or designee, patients with suboptimal response on at least 8 weeks of a steady dose of ruxolitinib may be allowed to de-escalate ruxolitinib therapy in order to enter a safety cohort which is enrolling patients at a lower dose; patients must receive the lower dose of ruxolitinib for at least 7 consecutive days without event before adding TGR-1202. If the patient completed screening evaluations including bone marrow biopsy/aspirate prior to ruxolitinib de-escalation, it need not be repeated after de-escalation provided that all evaluations occurred within 28 days prior to the first dose of TGR-1202.
* For expansion,

  * subjects may have a pathologically confirmed diagnosis of MF or PV as noted above in #2. There are also two expansion cohorts for patients with MDS/MPN (CMML, aCML, RARS-T or MDS/MPN-U) which warrants treatment. Patients with these diagnoses may be eligible, provided they are able to obtain ruxolitinib from commercial supply.
  * patients who have not yet received therapy with any JAK-STAT inhibitory agents or patients on at least 8 weeks of a steady dose of ruxolitinib; patients with exposure to other JAK-STAT inhibitory agents are not eligible.
* A bone marrow biopsy must be performed within four weeks prior to Cycle 1 Day 1 treatment to establish the baseline fibrosis score, and consent is required prior to that bone marrow biopsy to assure tissue is collected for protocol mandated testing;
* Subjects must have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2;
* Life expectancy of at least six months;
* Recovery to ≤ Grade 1 or baseline of any toxicities due to prior systemic treatments, excluding alopecia and anemia/thrombocytopenia assessed to be related to Ruxolitinib exposure;
* Women of child bearing potential (WCBP), defined as a sexually mature woman not surgically sterilized or not post-menopausal for at least 24 consecutive months if ≤55 years or 12 months if >55 years, must have a negative serum pregnancy test within 72 hours prior to the first dose of study drug and must agree to use highly effective methods of birth control throughout the study. Highly effective methods of contraception include total abstinence, sterilization of patient and/or patient's partner, or use of combination of two methods, including barrier methods (double barrier method is acceptable), IUD or IUS, and hormonal implants or combined oral contraceptives
* Must have adequate organ function as demonstrated by the following:
* ALT (SGPT) and/or AST (SGOT) ≤ 3x upper limit of normal (ULN), or ≤ 4 x ULN (if upon judgment of the treating physician, it is believed to be due to extramedullary hematopoiesis [EMH] related to MF); Total bilirubin ≤ 1.5 x ULN; or ≤ 2x ULN (if upon judgment of the treating physician, it is believed to be due to EMH related to MF); Serum creatinine ≤ 2.5 mg/dL x ULN; Hgb ≥ 8 g/dL; Plt ≥ 30k; ANC ≥ 750/uL

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from trial entry:

* Other invasive malignancies within the last 2 years, except non-melanoma skin cancer and localized cured prostate, cervical cancer, and DCIS
* History of cerebral vascular accident, unstable angina, myocardial infarction, or ventricular arrhythmia within the last 6 months;
* Any serious, unstable medical or psychiatric condition that would prevent, (as judged by the Investigator) the subject properly providing informed consent or any condition which would jeopardize compliance with the protocol
* Known history of human immunodeficiency virus (HIV), or known active hepatitis A, B, or C infection (hepatitis B carriers with normal LFTs and undetectable viral loads are allowed);
* Organ transplant recipients other than bone marrow transplant;
* Women who are pregnant or lactating;
* Autologous hematologic stem cell transplant within 3 months of study entry. Allogeneic stem cell transplant within 6 months. Grade II, or greater, active graft versus-host disease.
* Use of an investigational drug within 21 days or 5 half-lives (whichever is shorter) prior to the first dose of TGR-1202. For investigational drugs for which 5 half-lives is less than 21 days, a minimum of 10 days between termination of the investigational drug and administration of TGR-1202 is required.
* Previous therapy with GS-1101 (CAL-101), IPI-145 or any drug that specifically inhibits PI3K or mTOR within last 6 months;
* Any major surgery, chemotherapy, or immunotherapy within the last 21 days (limited palliative radiation is allowed ≥ 2 weeks); concurrent hydroxyurea is allowed if less than 2 grams daily and on stable dose for ≥14 days prior to study entry;
* Patient has received wide field radiotherapy (including therapeutic radioisotopes such as strontium 89) ≤ 28 days or limited field radiation for palliation ≤ 14 days prior to starting trial medications or has not recovered from side effects of such therapy;
* Ongoing immunosuppressive therapy (prednisone or equivalent ≤10 mg daily allowed as clinically warranted). Patients are allowed to use topical or inhaled corticosteroids;
* Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol
* Concurrent condition that in the investigator's opinion would jeopardize compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2023-03-21 (Actual); Study Completion 2024-05 (Actual)

PRIMARY OUTCOMES:
Safety of TGR1202 in combination with ruxolitinib | </=12 months
  All patients who have received at least one dose of TGR-1202 will be included in the safety population. All clinical safety data (vital signs, routine laboratory tests, and adverse events) will be tabulated and listed. The safety and tolerability of TGR-1202 and ruxolitinib will be evaluated by means of drug-related dose limiting toxicity, adverse event (AE) reports, physical examinations and laboratory safety evaluations.

SECONDARY OUTCOMES:
Overall response | EOT - 12 months
  Number of patients in each response category, polycythemia IWG response criteria, IWG-MRT response criteria, IWG MDS/MPN response criteria summarized as follows for target lesion criteria (see IWG for additional details): complete response (CR), normalization of bone marrow, peripheral counts, spleen size, and symptoms; partial response (PR); Hematologic improvement (HI), or progressive disease (PD). Patients are categorized according to the best response achieved prior to occurrence of progressive disease, where best response hierarchy is CR>PR>HI>SD>PD.
Total symptom score (MPN-TSS) | 16 weeks of therapy
  The myeloproliferative neoplasm - total symptoms score (MPN-TSS) is a validated tool in measurement in symptoms for patients with these diseases and we will measure patient reported outcomes with this validated tool
Blood levels of TGR1202 in combination with ruxolitinib (Pharmacokinetics) | 30 days
  The PK parameters (including AUC (0-∞), AUC (0- τ), Cmax, tmax, λz, and t½) of TGR-1202 and ruxolitinib following will be assessed by analysis of TGR-1202 plasma concentrations during the dose escalation phase of the study.

OTHER OUTCOMES:
TGR-1202's effects plasma cytokine levels when added to ruxolitinib | 0-16 weeks
JAK2V617F allele burden | 0-16 weeks
  Measurement of JAK2V617F allele burden by PCR
Mutations found on next generation sequencing (NGS) correlated with response | EOT 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Michael Savona, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (5):
- United States (5):
  - Mayo Clinic - Arizona, Phoenix, Arizona
  - University of Colorado Cancer Center, Aurora, Colorado
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Mays Cancer Center at University of Texas Health San Antonio, San Antonio, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://vicc.org/ct/